CLINICAL TRIAL: NCT03168971
Title: Managing Anxiety From Cancer (MAC): A Pilot Randomized Controlled Trial of a Psychological Intervention for Anxiety in Older Adults With Cancer and Their Caregivers
Brief Title: Managing Anxiety From Cancer (MAC): Testing an Intervention for Anxiety in Older Adults With Cancer and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-542; 5K23AG048632 (NIH)
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Depression; Quality of Life
Keywords: Cancer; Anxiety; Cognitive behavior therapy; Elderly; Caregivers; 18-542
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms

STUDY DESIGN:
Intervention Model Description: Patient-caregiver dyads will be randomly assigned to the intervention or a usual care control condition.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Managing Anxiety from Cancer (MAC) (Experimental): Older adults with cancer and their primary informal caregiver will receive a seven-session cognitive-behavior therapy intervention administered over the telephone by a trained study interventionist. The intervention is administered weekly and each session is 45-50 minutes in length. Patients and caregivers will receive the intervention independently and from separate therapists.
  Interventions: Behavioral: Managing Anxiety from Cancer (MAC)
- Usual Care (No Intervention): Older adults with cancer and their primary informal caregiver will receive standard care provided by their medical team. These participants will not receive any intervention from the research team.

INTERVENTIONS:
Behavioral: Managing Anxiety from Cancer (MAC) — The intervention consists of seven telephone-administered sessions. Session topics include psychoeducation on anxiety, behavioral strategies for managing anxiety, cognitive restructuring, communication skills training, acceptance techniques, problem-solving strategies, and planning for future anxiety. Session content is tailored for older adults and caregivers of older adults with cancer.
  Arms: Managing Anxiety from Cancer (MAC)

SUMMARY:
This study is being done to test the effects of Managing Anxiety from Cancer (MAC) therapy on anxiety compared to usual care, in patients and their caregivers. MAC is different from usual care because it uses a plan for managing anxiety that has been shown to work in previous studies. MAC has designed this plan for people 65 years of age and older. MAC also includes the primary caregiver which has been shown to help patients manage their anxiety.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS:

* Age 65 or older
* Confirmed diagnosis of breast, lymphoma, genitourinary, thoracic, gynecological or gastrointestinal cancer, currently on active treatment or within six months of completion of treatment
* As determined by the patient's primary oncologist and/or study staff, physically and cognitively able to complete study procedures
* English fluent (as per self-reported fluency of "very well")**
* In the judgment of the investigators and/or consenting professional, able to perform informed consent
* Has a primary informal caregiver (as defined by an unpaid individual who provides the patient with emotional, physical, and/or practical support) who is willing and able to participate in the study
* As part of the patient-caregiver dyad, at least one member reports elevated anxiety as defined by a score of 8 or greater on the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS)
* As per self-report, residency in New York or ability to complete sessions in New York
* Able to communicate over the phone for sessions
* Willingness to be audio-recorded for assessments and, if applicable, study sessions

CAREGIVERS:

* Age 21 or older
* In the judgment of the investigators and/or consenting professional, able to perform informed consent
* As part of the patient-caregiver dyad, at least one member reports elevated anxiety as defined by a score of 8 or greater on the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS)
* English fluent (as per self-reported fluency of "very well")**
* Is a primary informal caregiver (as defined by an unpaid individual who provides the patient with emotional, physical, and/or practical support) for an MSK patient
* As per self-report, residency in New York or ability to complete sessions in New York
* Able to communicate over the phone for sessions
* Willingness to be audio-recorded for assessments and, if applicable, study sessions

Exclusion Criteria:

PATIENTS:

* Endorsing active suicidal ideation on the item, "In light of your current circumstances, have you ever had thoughts of killing yourself?"
* As per oncologist or self-report, too weak or cognitively impaired to participate in the intervention and complete the assessments
* Per self-report/screening measures, has received cognitive-behavioral therapy since cancer diagnosis
* As per medical record or self-report, currently being treated for schizophrenia, substance use or dependence, and/or bi-polar disorder
* Anxiety due solely to a medical procedure as determined by a patient-report item on the screening questionnaire

CAREGIVERS:

* Endorsing active suicidal ideation on the item, "In light of your current circumstances, have you ever had thoughts of killing yourself?"
* Per self-report/screening measures, has received cognitive-behavioral therapy since patient"s cancer diagnosis
* As per self-report, currently being treated for schizophrenia, substance use or dependence, and/or bi-polar disorder
* If female, currently pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Anxiety sub-scale of the Hospital Anxiety and Depression Scale | Baseline (1-2 weeks after enrollment) and Follow-up (7-9 weeks after baseline)
  Change in anxiety from baseline to follow-up
Hamilton Anxiety Rating Scale | Baseline (1-2 weeks after enrollment) and Follow-up (7-9 weeks after baseline)
  Change in anxiety from baseline to follow-up

SECONDARY OUTCOMES:
Depression sub-scale of the Hospital Anxiety and Depression Scale | Baseline (1-2 weeks after enrollment) and Follow-up (7-9 weeks after baseline)
  Change in depression from baseline to follow-up
Distress Thermometer | Baseline (1-2 weeks after enrollment) and Follow-up (7-9 weeks after baseline)
  Change in distress from baseline to follow-up
Functional Assessment of Cancer Therapy-General: Emotional Quality of Life Sub-Scale (patients only) | Baseline (1-2 weeks after enrollment) and Follow-up (7-9 weeks after baseline)
  Change in health-related quality of life
Caregiver Quality of Life-Cancer (caregivers only) | Baseline (1-2 weeks after enrollment) and Follow-up (7-9 weeks after baseline)
  Change in health-related quality of life
Montgomery-Asberg Depression Scale | Baseline (1-2 weeks after enrollment) and Follow-up (7-9 weeks after baseline)
  Change in depression from baseline to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Trevino, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org